CLINICAL TRIAL: NCT06876324
Title: Adolescent SPEAKS Study: Integrating Supports to Promote PrEP for Black Adolescents Working With Apps
Brief Title: Integrating Supports to Promote PrEP for Black Adolescents Working With Apps
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Samantha Hill, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007320; 7K23MH128128-03 (NIH)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: HIV
Keywords: Medication Adherence; PrEP
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: AYAs will be paired with an adult who has identified as a support person and will use the app to facilitate dyadic communication to improve PrEP use among Black AYAs. Participants will be enrolled for 6 months. All participants will participate in the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AYA group (Experimental): All enrolled participants (AYAs and support persons) will receive a demonstration of the app including all of its features. All participants will use the app for 6 months. Each dyad of participants will instructed to use the app to communicate with each other and AYAs will be instructed to use the app to keep track of their PrEP. Data from the medication tracker will be collected at 1-, 3-, and 6-months
  Interventions: Behavioral: HealthMPowerment App

INTERVENTIONS:
Behavioral: HealthMPowerment App — A mobile health app designed to facilitate increased PrEP use and adherence among AYAs

SUMMARY:
This study applies Social Cognitive Theory to develop behavioral interventions promoting PrEP adherence. It seeks to adapt and test the enhanced HMP app for feasibility and acceptability among Black adolescents and young adults (AYAs) and adult supports.

DETAILED DESCRIPTION:
HIV pre-exposure prophylaxis (PrEP) is highly effective in preventing HIV infections, reducing the risk by over 90%. However, adherence among AYAs remains suboptimal, with only 34% maintaining adherence at 48 weeks. Studies suggest that adult support can improve adherence in pediatric HIV treatment, but this approach has not been systematically evaluated for PrEP use in AYAs. Prior research indicates that Black AYAs and their families are open to incorporating adult support for PrEP adherence.

Given the success of mobile health (mHealth) interventions in promoting sexual health, this study aims to enhance the HealthMPowerment (HMP) app-an existing mHealth platform designed for HIV prevention-to facilitate dyadic communication between Black AYAs and trusted adult support persons.

The study addresses the high rates of HIV among Black adolescents and young adults (AYAs) in Alabama, where AYAs (ages 13-24) account for 31% of new HIV diagnoses, with Black gay and bisexual males, transgender individuals, and heterosexual young women being disproportionately affected. Nearly half of new infections occur in rural areas. The U.S. Department of Health and Human Services Ending the HIV Epidemic initiative prioritizes Alabama as a geographic hotspot, emphasizing the need for patient-centered interventions to reduce HIV incidence.

ELIGIBILITY:
Inclusion Criteria:

* African Americans
* Living in the state of Alabama
* Have a PrEP indication (e.g. sex with a partner living with HIV, condomless sex, sex with multiple partners, engagement in transactional sex, or at least one sexually transmitted infection in the past 6 months)
* Support Person:

  * >21 years old
  * self-reported provision of instrumental, informational, or emotional support for a Black AYA 14-21 years old

Exclusion Criteria:

* HIV positive
* Inability to provide informed consent

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability/Usability | 1 month, 3 months, and 6 months
  The study evaluates an app's impact through post-intervention interviews, focusing on user experience, ethical concerns, and future usage intentions. It explores burden, satisfaction, attitudes, and how the app influences communication and adherence. Sekhon's Theoretical Framework of Acceptability will be utilized to measure this outcome.
Feasibility: Communication | 1 month, 3 months, and 6 months
  Communication between adolescents and young adults (AYA) and support person (i.e., Experience using chat features; Experience using forums). A modified version of Structured Assessment of FEasibility (SAFE) will be utilized to measure this outcome.

SECONDARY OUTCOMES:
Medication Adherence Tracker | 1 month, 3 months, and 6 months
  This will be measured by analyzing the percent of dates with data entered into the medication tracker and correlating that data with reasons why participants did not take their medication (when applicable)
Data Usage | 1 month, 3 months, and 6 months
  This will be measured by comparing the amount of time (minutes) spent using distinct features of the app (e.g. forums, educational resources, avatars, side effect trackers, chat features)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Hill, MD, MPH, Principal Investigator — Emory University
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Proposals should be directed to svhill2@emory.edu. To gain access, data requestors will need to sign a data access agreement. Data are delivered electronically to investigators.